CLINICAL TRIAL: NCT06790745
Title: Plasma Rich Fibrin Epidural Injection by Racz Catheter Versus Epidural Blood Patch in Postdural Puncture Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR939/11/24
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Plasma Rich Fibrin; Epidural; Racz Catheter; Epidural Blood Patch; Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Blood Patch, Epidural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural blood patch group (Experimental): Patients will receive epidural blood patch injection
  Interventions: Procedure: Epidural blood patch
- Plasma rich fibrin epidural injection by Racz catheter group (Experimental): Patients will receive plasma-rich fibrin epidural injection by Racz catheter
  Interventions: Drug: Plasma rich fibrin epidural injection by Racz catheter

INTERVENTIONS:
Procedure: Epidural blood patch — Patients will receive epidural blood patch injection
  Arms: Epidural blood patch group
Drug: Plasma rich fibrin epidural injection by Racz catheter — Patients will receive plasma rich fibrin injection by Racz catheter
  Arms: Plasma rich fibrin epidural injection by Racz catheter group

SUMMARY:
This study aims to evaluate plasma-rich fibrin epidural injection by Racz catheter and epidural blood patch in Post dural puncture headache.

DETAILED DESCRIPTION:
Post-dural puncture headache (PDPH) is also known as post-lumbar puncture (LP). PDPH is a major complication of neuraxial anesthesia that can occur following spinal anesthesia and with inadvertent dural puncture during epidural anesthesia.

Traditional management strategies include conservative measures such as oral analgesia, bed rest, oral or intravenous hydration, oral or intravenous caffeine, and administration of epidural crystalloid before catheter removal, but in refractory cases, more invasive techniques may be necessary. An epidural blood patch (EBP) has been the most favorable treatment for PDPH after an accidental dural puncture.

One innovative approach is the use of plasma-rich fibrin (PRF) derived from autologous whole blood, which contains and releases several different growth factors and cytokines to stimulate the healing of bone and soft tissue via degranulation. This approach has recently gained popularity in pain management. Another is the Racz catheter, a thin and flexible catheter used for targeted delivery of therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* Patients suffering from post-dural puncture headache.

Exclusion Criteria:

* Uncooperative patients.
* Severe comorbid conditions.
* Pregnancy.
* Anticoagulant therapy.
* Known allergies to plasma-rich fibrin or epidural blood patch components.
* Body mass index (BMI) ≥35 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Success rate of the procedures | 24 hours postoperatively
  The success rate of techniques for the treatment of headaches and associated symptoms on a 4-point rating scale (0 = none, 1 = slight, 2 = marked, 3 = complete relief) will be recorded.

SECONDARY OUTCOMES:
Degree of pain | 8 days postoperatively
  The degree of pain will be assessed using the Numeric Rating Scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at (0, 6, 12, 24, 48) h, 3, 4, 5, 6, 7, 8 days postoperatively.
Length of bed rest | 8 days postoperatively
  Length of bed rest after techniques and the efﬁcacy of techniques for the treatment of headaches and associated symptoms on a 4-point rating scale (0 = none, 1 = slight, 2 = marked, 3 = complete relief) will be recorded.
Change in optic nerve sheath diameter (ONSD) | 6 hours the procedure
  Optic nerve sheath diameter (ONSD) will be measured before and after 6 hours of the procedure.
Incidence of complications | 8 days postoperatively
  Incidence of complications that may occur during the technique such as (bending of the tip of the needle, shearing of the catheter, misplacement of the catheter, blocking of the catheter, blood aspiration and bleeding in the epidural space, hypotension, migration of the catheter, paresthesia, headache and infection) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author